CLINICAL TRIAL: NCT04888286
Title: Donor-specific Anti-HLA Antibodies (DSAS) in Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation From Mismatched Donors
Brief Title: DSAs in Patients Undergoing Allo-HSCT From Mismatched Donors
Acronym: AIBT_DSAs
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano Trapianto di Midollo Osseo (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Sponsor
Other Study IDs: GITMO-AIBT DSAs
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Hematologic Diseases; Stem Cell Transplant Complications
Keywords: Retrospective survey; GITMO; Hematological disease; Allogeneic stem cell transplantation; anti-HLA antibodies; mismatched donors; DSAs searching
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients who underwent mismatched allogeneic transplantation: Pediatric and adult patients who underwent mismatched allogeneic transplantation, from January 2014 to June 2017.

SUMMARY:
Retrospective observational multicentric, spontaneous non-interventional non-pharmacological Italian study. The primary objective is analysis of Anti-HLA antibodies and DSAs searching and monitoring activities in haematological adult and paediatric patients undergoing allo-HSCT from January 2014 to June 2017. This study will evaluate approximately 1000 subjects (with competitive enrolment) from GITMO investigational centers.

DETAILED DESCRIPTION:
The aim of the study is to evaluate, retrospectively, the activity of the Italian Centres in the search for donor-specific anti-HLA antibodies (DSAs) in patients undergoing allogeneic hematopoietic stem cell transplantation from mismatched donors and the strategy of treatment employed in case of DSAs positivity. Moreover, the study aims are to evaluate the role of DSAs on the engraftment. The interest in the study arises from the absence of knowledge on the MFI cut-off value clinically significant, and from the absence of the knowledge on the role of DSAs against each HLA locus on the engraftment and post-transplant survival. Furthermore, shared desensitization protocols and common donor selection strategies are lacking.

In recent years, with the increase of haploidentical and mismatched unrelated donor transplants, is also increasing the interest for DSAs at the time of HSCT, considering their potential role on graft failure by cell-mediated or antibody-mediated mechanisms.

Having a picture of the policy about DSAs management in Italian Transplant Centers, and of the indications reported by the Histocompatibility and Immunogenetic Laboratories, will allow to define, in collaboration with GITMO / AIBT, a consensus strategy. This strategy could be the platform for prospective studies.

The study involves the enrolment of patients (adults and paediatrics) undergoing mismatched allogeneic transplant, in the period 2014-2017 regardless of the source of stem cells and the search for DSAs. The sample size includes all the transplants recorded in the Gruppo Italiano Trapianti di Midollo Osseo and European group for Blood and Marrow Transplantation database.

Primary objectives are two: the analysis of Anti-HLA antibodies and DSAs searching and monitoring activities in haematological patients undergoing Allogeneic Hematopoietic Stem Cell Transplantation (HSCT) performed by Histocompatibility and Immunogenetic Laboratories in collaboration with Italian transplant centres and assess to the impact of DSAs on neutrophil and platelet engraftment.

The secondary objectives are to study the probability and times to neutrophils and platelets engraftment, reject, poor engraftment in patients undergoing HSCT among different transplant centres, according to anti-HLA antibodies and DSA testing practice and assess the Overall Survival (OS) in patients undergoing HSCT with or without DSAs.

The analysis of continuous and categorical variables will be performed according to the criteria of descriptive statistics, including mean, median, standard deviation, range, minimum and maximum values for continuous variables, absolute and relative values for categorical variables. For the comparison of continuous and categorical variables, parametric and non-parametric statistical tests (Chi-square test, Fisher exact test and rank correlation coefficient of Spearman) will be applied. Competitive risk analysis will be used to assess the cumulative incidence (CI) of engraftment, considering death within 60 days as a competitive event.

OS will be estimated according to the Kaplan-Meier method and calculated from the date of the transplant; the comparison between different groups will be performed with the log-rank test.

The Cox regression model for proportional hazards will be used for multivariate analysis in order to evaluate the prognostic effect of the various variables in terms of engraftment. For the statistical analysis, a p-value <0.05 will be considered statistically significant.

This trial is being organized under the auspices of the Gruppo Italiano Trapianti di Midollo Osseo that involves the principal Centres active in transplantation of any kind of hematopoietic stem cells (HSCT) in Italy.

The study will be conducted according to the principles of Good Clinical Practice, the current Italian and European laws and regulations, in agreement with the declaration of Helsinki. The protocol has been written and the study will be conducted according to The International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) Harmonized Tripartite Guideline for Good Clinical Practice, issued by the European Union. The responsible Local Ethical Committee approval must be obtained before starting the trial. A copy of the patient informed consent form must be submitted to the appropriate authority or committee, together with the protocol for written approval. Written approval of the protocol and informed consent by the responsible and appropriate authority or committee must be obtained prior to recruitment of patients to the study.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent mismatched allogeneic transplantation, from January 2014 to June 2017
* signed the informed consent

Exclusion Criteria:

* Absence of consent Written information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and children allogenic Hematopoietic stem cell transplantation recipients
Sampling Method: Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Analysis of the monitoring practice of DSAs | 6 months from allogeneic hematopoietic stem cell transplantation
  The variables that will be collected are: Type of transplant in which the search for DSAs is carried out, Laboratory methods used, Positivity cut-off used, Donor selection criteria if DSAs present, Desensitization protocol employed
Role of DSAs on neutrophils and platelets engraftment | 28 days from allogeneic hematopoietic stem cell transplantation
  Time to reach an absolute neutrophil count > 0.5 109/L from day of HSCT. Neutrophil recovery end-point will be defined as the first of 3 consecutive days with an absolute neutrophil count > 0.5 x109/L.
  Time engraftment of platelet count will be defined as PTLS >20.9 x 109/L without transfusion requirements for at least 5 days.
Graft failure | 28 days from allogeneic hematopoietic stem cell transplantation
  graft failure is defined as peripheral blood ANC < 0.5 × 109/L by after allogeneic hematopoietic stem cell transplantation without evidence of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Anna Paola Iori, Principal Investigator — Azienda Policlinico Umberto I
Locations (25):
- Italy (25):
  - Clinica di Ematologia. AOU Ospedali Riuniti di Ancona, Ancona
  - Policlinico di Bari-Ematologia con trapianti, Bari
  - Divisione di Ematologia - Ospedali Papa Giovanni XXIII, Bergamo
  - Ospedale Seragnoli Malpighi, Bologna
  - AO Spedali Civili di Brescia- USD - TMO Adulti, Brescia
  - S.C. Ematologia - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliera di Careggi, Florence
  - AOU IRCCS San Martino - IST, Genova
  - Ospedale Gaslini, Genova
  - Div. di Ematologia e TMO, Istituto Nazionale Tumori, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Unità Operativa di Ematologia e Trapianto Midollo Osseo (UTMO), Ospedale San Raffaele di Milano, Milan
  - Azienda ospedaliera Santobono Pausilipon, Napoli
  - Azienda ospedaliera Universitaria di Parma, Parma
  - Fondazione IRCCS San Matteo, Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Ospedale San Carlo, Potenza
  - Centro Unico Regionale Trapianti di Midollo Osseo - Ospedale Bianchi-Melacino-Morelli, Reggio Calabria
  - A.O. San Camillo Forlanini, Roma
  - Divisione di Ematologia - Istituto di Semeiotica Medica - Policlinico A. Gemelli, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I - Università La Sapienza, Roma
  - Azienda ospedaliera Città della Salute e della Scienza, Torino
  - Clinica Ematologica - AOU Santa Maria Della Misericordia, Udine
  - Policlinico GB Rossi, Verona